CLINICAL TRIAL: NCT03641287
Title: The Effects of Moderate Exercise on Distress, Quality of Life, and Biomarkers of Angiogenesis and Chronic Stress in Ovarian Cancer Survivors - A Randomized Controlled Trial
Brief Title: The Effects of Exercise on Distress, Quality of Life, and Biomarkers in Ovarian Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment ended early due to the funding timeline
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kathryn Pennington, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RG1001826; 10045 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2018-01630 (Registry Identifier: NCI / CTRP); R21CA215662 (NIH)
Record Dates: First submitted 2018-08-15; First posted 2018-08-22 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Cancer; Fallopian Tube Adenocarcinoma; Fallopian Tube Carcinosarcoma; Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; Malignant Ovarian Brenner Tumor; Ovarian Adenocarcinoma; Ovarian Carcinosarcoma; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Ovarian Undifferentiated Carcinoma; Primary Peritoneal Serous Adenocarcinoma; Primary Peritoneal Carcinosarcoma; Primary Peritoneal Transitional Cell Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Brenner Tumor | interventions — Exercise; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (aerobic exercise) (Experimental): Participants meet with exercise physiologist for 1, 60 minute session. Participants then receive individualized exercise prescription with goal of moderate aerobic exercise over 150 minutes per week at home for up to 24 weeks. Participants also receive telephone-based motivational support by exercise physiologist weekly for 24 weeks.
  Interventions: Other: Exercise Counseling; Other: Aerobic Exercise; Other: Physiological Support; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (habitual level of physical activity) (Active Comparator): Participants maintain habitual levels of physical activity and receive general education material about ovarian cancer and survivorship for 24 weeks. After 24 weeks, participants are offered exercise intervention.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Best Practice

INTERVENTIONS:
Other: Exercise Counseling — Meet with exercise physiology
  Arms: Arm I (aerobic exercise)
Other: Aerobic Exercise — Receive prescription for moderate aerobic exercise
  Other Names: Aerobic Activity, aerobic exercise
  Arms: Arm I (aerobic exercise)
Other: Physiological Support — Receive motivational support via telephone care
  Arms: Arm I (aerobic exercise)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Best Practice — Undergo habitual level of physical activity
  Other Names: best practice, standard of care, standard of care, standard therapy
  Arms: Arm II (habitual level of physical activity)

SUMMARY:
Many individuals with ovarian cancer experience distress, fatigue, weakness, anxiety, and other symptoms that decrease quality of life. Moderate exercise may improve quality of life, decrease distress, and improve biomarkers associated with prognosis in individuals with ovarian cancer. This clinical trial studies how well moderate exercise works in improving distress, quality of life, and biomarkers of angiogenesis and chronic stress in individuals with ovarian, fallopian tube, and primary peritoneal cancer.

DETAILED DESCRIPTION:
OUTLINE:

Patients are randomized to 1 of 2 arms.

ARM I (EXERCISE INTERVENTION): Patients meet with exercise physiologist for 1, 60 minute session. Patients then receive individualized exercise prescription with goal of moderate aerobic exercise over 150 minutes per week at home for up to 24 weeks. Patients also receive telephone-based motivational support by exercise physiologist weekly for 24 weeks.

ARM II (CONTROL GROUP): Patients maintain habitual levels of physical activity and receive general education material about ovarian cancer and survivorship for 24 weeks. After 24 weeks, patients are offered exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage II-IV epithelial ovarian, fallopian tube, or peritoneal cancer. If site of origin cannot be specified, carcinoma of Mullerian origin may be included if most consistent with ovarian/fallopian tube/peritoneal origin rather than uterine origin. The following histologic epithelial cell types are eligible: serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, clear cell carcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's tumor, undifferentiated carcinoma, carcinosarcoma, or adenocarcinoma not otherwise specified. Women with neoplasms of low malignant potential (borderline tumors) are not eligible.
* Subjects must have no evidence of disease, as defined by their treating oncologist, and with normal CA-125 (=< 35).
* Subjects must have completed primary surgery and adjuvant chemotherapy for treatment of ovarian, fallopian tube, of peritoneal cancer within one to six months of screening. Maintenance therapy will be allowed as long as the participant is in clinical remission- including hormonal agents, anti-angiogenesis agents, PARP inhibitors, and immunotherapy. Prior radiation therapy is allowed, as long as it has been completed within one to six months of screening. Subjects may have received prior therapies (including surgery, chemotherapy, radiation therapy) for other malignancies in the past.
* Eastern Cooperative Oncology Group (ECOG) status of 0, 1, or 2.
* Pregnancy and the need for contraception:

  * Participants with ovarian cancer have undergone hysterectomy with removal of ovaries and tubes as part of surgical treatment, and therefore do not have the potential to become pregnant.
* Ambulatory.
* Ability to understand and the willingness to sign a written informed consent document.
* Individuals participating in most other clinical trials are eligible provided their enrollment in the other trial does not impair their ability to participate in the physical activity interventions and study assessments required in this trial. The other clinical trial must not be a behavioral intervention trial.

Exclusion Criteria:

* Subjects who have had primary surgery, chemotherapy and/or radiation therapy within 4 weeks prior to screening. Subjects may have received other surgeries not performed for primary treatment (for example, removal of intraperitoneal port, laparoscopic cholecystectomy, etc.) within 1 month of screening as long as they do not have post-operative restrictions that would preclude participating in a moderate intensity exercise program once enrolled in the clinical trial.
* Self-reported inability to walk at least 2 blocks (at any pace).
* Prior brain metastasis is not an exclusion, as long as subject is in clinical remission.
* Uncontrolled or concurrent illness including, but not limited to: unstable angina pectoris, recent (within six months) myocardial infarction, uncontrolled cardiac arrhythmia, uncontrolled congestive heart failure, hypertrophic obstructive cardiomyopathy, uncontrolled hypertension (systolic > 200, diastolic > 120), conditions (cardiovascular, respiratory, or musculoskeletal disease or joint problems) that preclude moderate physical activity. Subjects with a history of cardiac arrest, or those with moderate/severe aortic or mitral stenosis may be eligible if their treating physician determines that moderate physical activity is safe. Moderate arthritis that does not preclude physical activity is not a reason for ineligibility. Individuals with lymphedema or peripheral neuropathy will not be excluded. They will be evaluated by the exercise physiologist for safety and modifications to the exercise prescription will be made as appropriate.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Already physically active > 90 minutes per week of moderate exercise.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Pennington, Principal Investigator — University of Washington
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Habitual Level of Physical Activity)
Started | 31 | 33
Completed | 28 | 33
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Habitual Level of Physical Activity) | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.77 (9.68) | 63.73 (10.69) | 62.78 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 64
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 27 | 31 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 28 | 26 | 54
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 33 | 64
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.73 (5.31) | 28.92 (7.17) | 27.86 (6.39)
Stage [Count of Participants; unit: Participants] — Cancer is staged as stage I, II, III, or IV using FIGO 2014 staging system. A higher stage is associated with worse prognosis.
  Participants
    Stage II | 3 | 4 | 7
    Stage III | 22 | 17 | 39
    Stage IV | 6 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life Measured Using the RAND 36-item Short Form Health Survey Physical Component Score
Description: Will be measured using the RAND 36-item Short Form Health Survey Physical Component Score. Mean change from baseline to 24 weeks between the exercise intervention and control group in the RAND 36-item Short Form Health Survey Physical Component Score.
  RAND 36-Item Short Form assesses eight subscales including physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, general health perceptions, and perceived change in health. Possible scores for each subscale range from 0 to 100. The Physical Component Score (PCS) is an aggregate of the eight subscales using a standardized algorithm, with a mean of 50 and standard deviation of 10 in the general US population. Possible scores range from 20 to 60, with higher scores indicating a better quality of life.
Time Frame: Baseline up to 24 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Habitual Level of Physical Activity)
Number analyzed (Participants) | 28 | 27
score on a scale | 4.37 (0.99) | 4.61 (2.02)

2. Primary Outcome: Change in Distress, Measured Using the Perceived Stress Scale
Description: Will be measured using the Perceived Stress Scale. Mean change from baseline to 24 weeks between the exercise intervention and control group in the Perceived Stress Scale.
  The Perceived Stress Scale is a 10 item questionnaire with a total score range of 0-40. Higher total scores indicate higher distress.
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Habitual Level of Physical Activity)
Number analyzed (Participants) | 28 | 28
score on a scale | -1.4 (0.97) | 1.05 (1.64)

3. Primary Outcome: Change in Distress, Measured Using the Hospital Anxiety and Depression Scale - Anxiety Subscale
Description: Will be measured using the Hospital Anxiety and Depression Scale - Anxiety subscale. Mean change from baseline to 24 weeks between the exercise intervention and control group in the Hospital Anxiety and Depression Scale - anxiety subscale.
  The Hospital Anxiety and Depression Scale includes 2 subscales: anxiety and depression.
  The Hospital Anxiety and Depression Scale - anxiety subscale total scores range from 0 to 21; higher scores indicated greater severity of anxiety symptoms.
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Habitual Level of Physical Activity)
Number analyzed (Participants) | 28 | 28
score on a scale | -1.15 (0.56) | -0.15 (0.72)

4. Primary Outcome: Change in Distress, Measured Using the Hospital Anxiety and Depression Scale - Depression Subscale
Description: Will be measured using the Hospital Anxiety and Depression Scale - Depression sub scale. Mean change from baseline to 24 weeks between the exercise intervention and control group in the Hospital Anxiety and Depression Scale - Depression subscale.
  The Hospital Anxiety and Depression Scale includes 2 subscales: anxiety and depression.
  The Hospital Anxiety and Depression Scale - Depression subscale total scores range from 0 to 21; higher scores indicated greater severity of depression symptoms.
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Habitual Level of Physical Activity)
Number analyzed (Participants) | 28 | 28
score on a scale | -0.76 (0.42) | -0.32 (0.80)

5. Primary Outcome: Change in IL-6 (Biomarker of Angiogenesis)
Description: Mean change from baseline to 24 weeks between the exercise intervention and control group in mean levels of IL-6.
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Habitual Level of Physical Activity)
Number analyzed (Participants) | 25 | 23
pg/mL | -0.57 (2.03) | 0.09 (0.54)

6. Primary Outcome: Change in VEGF (Biomarker of Angiogenesis)
Description: Mean change from baseline to 24 weeks between the exercise intervention and control group in mean levels of VEGF.
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Habitual Level of Physical Activity)
Number analyzed (Participants) | 25 | 23
pg/mL | -37.3 (41.84) | -82.2 (36.35)

7. Primary Outcome: Change in Nocturnal Cortisol (Biomarker of Chronic Stress)
Description: Mean change from baseline to 24 weeks between the exercise intervention and control group in mean level of evening salivary cortisol.
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Error); unit: ug/dL
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Habitual Level of Physical Activity)
Number analyzed (Participants) | 27 | 23
ug/dL | 0.01 (0.157) | 0.11 (0.07)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Habitual Level of Physical Activity)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33

LIMITATIONS AND CAVEATS:
Enrollment ended before meeting accrual goal due to the funding timeline, leading to smaller numbers of participants analyzed.

Most participants completed the study after the COVID-19 pandemic began. The study continued for several years during the pandemic. Multiple surges occurred and there was variable timing of infections experienced by participants and their loved ones over the course of their 6 month study participation. Participants were not uniformly affected by the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT03641287/Prot_SAP_000.pdf